CLINICAL TRIAL: NCT00024323
Title: A Phase I Study of 3-Aminopyridine-2-Carboxaldehyde Thiosemicarbazone (3-AP, Triapine) Administered Daily x 5 in Combination With Cisplatin
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: VION-CLI-021; CDR0000068918 (Registry Identifier: PDQ (Physician Data Query)); NCI-V01-1668
Record Dates: First submitted 2001-09-13; First posted 2003-06-20 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2002-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

INTERVENTIONS:
Drug: cisplatin
Drug: triapine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining 3-AP with cisplatin in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of cisplatin when administered with 3-AP in patients with advanced cancer.
* Determine the toxic effects of this regimen in these patients.
* Determine the antitumor responses in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of cisplatin.

Patients receive 3-AP IV over 2 hours on days 1-4 and cisplatin IV over 1 hour on days 2 and 3. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of cisplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 15-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed progressive malignant disease that has failed at least 1 conventional treatment or is unlikely to respond to current therapy
* Measurable or evaluable disease

  * Elevated serum tumor marker considered evaluable disease
* No known active CNS metastases

  * Previously treated CNS metastases with no evidence of new CNS metastases allowed if stable for at least 2 months

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL (transfusion allowed)
* No active bleeding or coagulation disorder (except occult blood related to gastrointestinal cancer)

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* ALT and AST no greater than 3 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 5 times ULN
* PT and PTT no greater than 1.5 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No active heart disease
* No myocardial infarction within the past 3 months
* No symptomatic coronary artery disease
* No uncontrolled arrhythmias
* No uncontrolled congestive heart failure

Pulmonary:

* No moderate to severe compromise of pulmonary function

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infectious process
* No pre-existing severe hearing impairment
* No grade 2 or greater neuropathy
* No other life threatening illness
* No prior severe allergic reaction to cisplatin
* No mental deficits and/or psychiatric history that would preclude study
* No persistent chronic toxic effects from prior chemotherapy greater than grade 1

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 2 weeks since prior biologic therapy

Chemotherapy:

* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* At least 3 months since prior cisplatin or platinum analogue
* No prior 3-AP

Endocrine therapy:

* At least 2 weeks since prior hormonal therapy

Radiotherapy:

* More than 3 weeks since prior radiotherapy

Surgery:

* At least 3 weeks since prior major surgery and recovered

Other:

* No other concurrent investigational drugs
* No other concurrent nephrotoxic drugs (e.g., aminoglycoside antibiotics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (2):
- United States (2):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Yale Comprehensive Cancer Center, New Haven, Connecticut

REFERENCES:
- [Derived] Kunos CA, Chu E, Beumer JH, Sznol M, Ivy SP. Phase I trial of daily triapine in combination with cisplatin chemotherapy for advanced-stage malignancies. Cancer Chemother Pharmacol. 2017 Jan;79(1):201-207. doi: 10.1007/s00280-016-3200-x. Epub 2016 Nov 22. PMID 27878356